CLINICAL TRIAL: NCT00491088
Title: The CPAP Effect in Severe Obstructive- Sleep- Apnea Patients Without Daytime Sleepiness: A Control Randomized Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Peilin Lee/attending physician, National Taiwan University Hospital
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 200701063R
Record Dates: First submitted 2007-06-21; First posted 2007-06-25 (Estimated); Last update posted 2010-03-01 (Estimated); Status verified 2010-02

CONDITIONS: Sleep Apnea, Obstructive
MeSH Terms: conditions — Sleep Apnea, Obstructive

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Device: CPAP — CPAP for 12 weeks

SUMMARY:
Specific Aim:

1. To prove our hypothesis that in severe OSA patients without daytime sleepiness, CPAP worked as effectively as in severe OSA patients with daytime sleepiness.

   Using sham CPAP as the optimal placebo, we conduct a randomized double-blind placebo controlled trial to assess the CPAP effect in severe OSA patients without daytime sleepiness.
2. To establish a model to predict the CPAP effect We use the parameters of five aspects, including changes of polysomnographic parameters, improvement of sleepiness, fatigue and QOL, sympathetic activity, inflammatory mediators and metabolism, to establish a model to predict CPAP effect.

DETAILED DESCRIPTION:
Obstructive sleep apnea (OSA) is a common disease, which affects 4% middle-aged men and 2% women. Daytime sleepiness is one of the symptoms of OSA which drive patients to seek medical help. Sleepiness in OSA has been reported to be raised by microarousal, altered sleep structure and somnogenic cytokine and modifications in body metabolism. The assessments of daytime sleepiness included objective measures, like multiple sleep latency test and subjective measures, like Epworth sleepiness scale (ESS).

So far, continuous positive airway pressure (CPAP) is the standard treatment for patients with severe OSA. CPAP could improve daytime wakefulness, blood pressure and quality of life (QOL). Several studies tried to identify factors predicting the CPAP effect and most concluded CPAP was not effective for patients with high apnea-hypopnea index but not sleepy. All of them determine the CPAP effect in terms of daytime function, lowering of blood pressure and QOL. None of these studies evaluate the CPAP effects in terms of improvement of sympathetic hyperactivity, inflammatory mediators and metabolic abnormalities. Therefore, we assumed patients whose daytime functions didn't improve after CPAP treatment still possibly got benefit from altering factors contributing to cardiovascular consequences.

Our previous study showed that CPAP effect in OSA patients without sleepiness was as well as in patients with sleepiness, except that plasma level of norepinephrine and 24hr mean arterial blood pressure could be lowered more in patients with sleepiness. However, without optimal placebo and randomization, the actual role of CPAP in treating non-sleepy OSA patients still couldn't be determined.

Recently sham CPAP was developed, which mimicked all the characteristics of a true CPAP except for the null pressure applied to the upper airway of the patient. Moreover, sham CPAP doesn't influence sleep efficiency, arousals, or apnea-hypopnea index. Therefore, in this project, using sham CPAP as a placebo, we propose a randomized double-blind placebo controlled trial to assess the effectiveness of CPAP in severe OSA patients without daytime sleepiness. We also establish a model to predict the CPAP effect. The results would change the current practice of managing severe OSA patients without daytime sleepiness.

ELIGIBILITY:
Inclusion Criteria:

* Severe obstructive sleep apnea (AHI>=30/hr) age, sex, BMI match control subject

Exclusion Criteria:

Patients were excluded when they:

* Refused to participate in this study
* Had severe obstructive pulmonary disease or active neurological events
* Enrolled in other studies at the same time

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Estimated)
Dates: Start 2007-06; Primary Completion 2009-08 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
improvement of sleepiness | after 4-week and 12-week CPAP treatment

SECONDARY OUTCOMES:
improvement of fatigue and QOL, sympathetic activity, inflammatory mediators and metabolism | after 4-week and 12-week CPAP treatment

CONTACTS AND LOCATIONS:
Overall Officials: Whey Dong Wu, M.D., Principal Investigator — National Taiwan University Hospital; Peilin Lee, M.D., Principal Investigator — National Taiwan University Hospital
Locations (1):
- Naitonal Taiwan University Hospital, Taipei, Taiwan